CLINICAL TRIAL: NCT02409147
Title: Initiation of a Deceased Donor Uterine Transplantation Program at the University of Nebraska Medical Center
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0138-15-FB
Record Dates: First submitted 2015-03-27; First posted 2015-04-06 (Estimated); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Uterus Transplant
MeSH Terms: interventions — thymoglobulin; Basiliximab; Tacrolimus; Mycophenolic Acid; Prednisone; Trimethoprim, Sulfamethoxazole Drug Combination; Valganciclovir; Aspirin; Nystatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Healthy female volunteers wishing to have a childbirth via uterine transplantation
  Interventions: Procedure: Uterine Transplant

INTERVENTIONS:
Procedure: Uterine Transplant — Surgical implantation of a deceased donor uterus, induction therapy with thymoglobulin or basiliximab, maintenance immunosuppression with Prograf, Cellcept, and Prednisone. Anti-infective treatment with Bactrim and Valcyte and Nystatin. Anti-platelet therapy with aspirin. IVF per standard protocol. At time of birth: ceasarean section. Ultimately, transplant hysterectomy.
  Other Names: Thymoglobulin; Basiliximab; Prograf; Cellcept; Prednisone; Bactrim; Valcyte; Aspirin; Nystatin

SUMMARY:
This study will explore the feasibility of initiating a uterine transplant program at UNMC. Using the procedural templates established by a successful Swedish team, the investigators will identify emotionally and socially stable females of reproductive age with intact ovaries who are unable to gestate a child due to congenital or acquired uterine factor infertility (UFI). Women will be 21 to 35 years of age upon entry into the protocol, with normal ovarian reserve and otherwise healthy for pregnancy. After careful screening, participants will undergo egg harvest, in-vitro fertilization, and embryo cryopreservation using standard methods. Women who successfully complete in vitro fertilization and cryopreservation of at least six embryos will be eligible to receive implantation of a deceased donor uterus. After a period of observation to ensure normal menstrual cycling and graft viability, embryo implantation will be undertaken. Gestations will be carefully monitored by our high-risk pregnancy specialists. Medical research interventions include uterine harvest from a deceased donor, surgical implantation of the organ utilizing standard transplant techniques, careful post-transplant follow-up including immune suppression therapy tailored to minimize fetal compromise, and careful management of pregnancy. After childbearing is complete (at most two gestations), the donor uterus will be removed. In addition, open-ended interviews and written surveys will be conducted to elicit ethical and psychosocial concerns arising from the experience of subjects and their families, health care providers, and the wider community. The investigators intent is to monitor outcomes lifelong for transplant recipients and live-born infants.

DETAILED DESCRIPTION:
Uterine transplantation was developed as a surgical/medical procedure to ameliorate the condition of absolute uterine factor infertility. As a condition, the congenital or acquired state renders fertile-age women the inability to have a child via conventional birth. It is estimated that this condition may affect near 1 in 500 women. The alternative, namely gestational surrogacy or adoption, can be fraught with legal, ethical, or religious issues. Significant research and progress has been obtained in Europe (namely Sweden) in facilitating uterine transplantation. Recently, they were able to obtain a successful live childbirth using a donated uterus from a living relative. Based on significant background research already performed, the aim of this research study is to expand upon their gains by successfully establishing a deceased donor uterus transplantation program at UNMC.

Prior to the success of the Swedish team, two other European/Asian medical research groups have attempted deceased donor uterus transplantation. The first resulted in organ failure from unclear pathology. The second was a successful transplant, but failed to yield a childbirth due to multiple miscarriages. In 2004 however, the team from the Sahlgrenska Institute in Gothenburg instituted a rigorous research undertaking in order to study the phenomenon and to obtain a childbirth. Using established immunological knowledge, and practical experience using animal models, the investigators were able over a course of a decade, to start an active transplant program.

From a medical/obstetrics and gynecology standpoint, potential subjects were screened using a rigorous physical and psychosocial evaluation. This involved meeting with multiple members of the research team, in addition to independent monitors familiar with the field and the risks and benefits of participation. To facilitate success, all women and their partners underwent investigation to rule out any sterility factors that could have been related to fertility. Next, egg harvesting and embryo transfer was undertaken according to currently accepted protocols. Of note, all women who had uterine agenesis had some type of neo-vaginal recreation in order to facilitate IVF. Finally, donor and recipient HLA matching was done using standard transplantation methods in order to avoid unacceptable matches.

During surgery, the donor underwent an extensive procedure in order to successfully dissect out the artery and venous supply of the organ. The vagina was transected caudal to the fornix, thus allowing a donor specimen which was attached by only the vascular pedicles. (The process of removing a uterus from a living donor is infinitely more complex than that of a deceased donor, hence our initial plan at UNMC is to focus on organs derived from the latter.) Once the organ was removed, it was flushed with preservation solution using standard transplantation protocols. The recipient surgery was also performed in standard fashion, with the donor iliac vessels anastomosed to the recipients. The vaginal rim of the graft was sutured to the recipient's vagina in standard fashion. Routine intra-operative examinations with Doppler (to assess blood flow) were then performed prior to the termination of the operation.

Maintenance immunosuppression was given to the recipients using standard accepted protocols with close monitoring of drug levels. Serial Doppler US were done both during hospitalization and in follow up to assess uterine viability. Clinical examination from an obstetrician was performed at pre-determined intervals and biopsies of uterine tissue were taken to assess for organ viability and to rule out rejection. Those few patients who did have rejection were treated with standard transplantation protocols with increased steroids only.

Embryo transfer was done at approximately 1 year post transplant, in order to ensure continued viability and normal menstruation of the organ. Post transfer, hormonal stimulation was done using standard reproductive endocrinology protocols. Serial monitoring of the fetus was done at routine intervals through the 9 month gestational period. Finally, a caesarean section was performed in routine fashion at time of birth.

Our groups rationale at UNMC is to continue to build on the accepted protocols developed by the Swedish team and apply them to deceased donors. The investigators believe our vast experience in transplant and obstetrics/gynecology combined with reproductive endocrinology facilitates undergoing this exciting new medical and surgical therapy.

ELIGIBILITY:
Inclusion Criteria:

* For transplantation, the criteria are as follows:

  1. Female of reproductive age with intact native ovaries and no medical contraindication to transplantation, including surgical procedure and subsequent immunosuppression, and no medical contraindication to reproduction and gestation in a transplanted uterus. Evaluation for a medical contraindication will be determined by a maternal-fetal medicine specialist at UNMC.
  2. Diagnosed with either congenital or acquired uterine factor infertility (UFI) and counseled about alternate options for family building including gestational surrogacy and/or adoption and provided access to these alternate services. Acquired circumstances may include nonfunctional uterus and hysterectomy due to benign disease (uterine fibroids, Asherman's syndrome, pelvic infection, postpartum hemorrhage) or gynecologic malignancy of the uterus or cervix. Additionally, UFI may be a result of congenital anomaly of the uterus and uterine agenesis.
  3. If uterine removal was for uterine or cervical cancer a minimum 5 year recurrence-free time period will be required.
  4. If MRKH Syndrome (Mayer-Rokitansky-Kuster-Hauser) or Mullerian agenesis is present, the patient has a negative evaluation for other relevant congenital abnormalities (such as a pelvic kidney). Additionally, women with Mulllerian agenesis who have absence of the vagina must have had neovaginal creation surgery prior to uterine transplant in order to allow for embryo transplantation and monitoring of the organ after transplant.
  5. Ovaries are intact with adequate ovarian reserve as determined by accepted markers including anti-Mullerian hormone level (AMH), astral follicle count and/or early follicular follicle stimulating hormone (FSH) levels.
  6. Desires a biological child and is unable or unwilling to consider gestational surrogacy, and / or seeks uterine transplantation as a means to experience gestation, with an understanding of the limitations provided by the uterine transplant in this respect.
  7. Meets psychological evaluation criteria, e.g.,stable, committed relationship with an individual who supports uterine transplant and intends to co-parent; emotionally mature with good coping skills and no significantly adverse mental health history; normal intellect allowing careful analysis of risks and benefits; no evidence of coercion; no significant evidence of previous noncompliance with medical care; no evidence of frank unsuitability for motherhood (e.g., previous conviction for child abuse).
  8. Likely to comply with medical management, including antirejection immune suppression, frequent follow-up with surgical team, time-sensitive reproductive endocrinology management, high-risk pregnancy management, possible high-risk neonatal management.
  9. Likely to be able to accommodate potential adverse outcomes such as loss of graft, inability to conceive, loss of pregnancy, adverse fetal or neonatal outcome.
  10. Willing to consider transplant hysterectomy or termination of pregnancy if medically necessary.
  11. Willing to undergo oocyte harvest and in-vitro fertilization prior to transplantation, with at least six viable embryos cryopreserved in anticipation of post-transplant implantation.
  12. Financially able to cover anticipated expenses of assisted reproductive services, either through third party coverage or through personal assets.

Exclusion Criteria:

* For transplantation: Exclusions include genetic males, and women who do not meet the inclusionary criteria above. Residence in the greater Omaha area during the implantation and pregnancy period is required because of the time-sensitive nature of transplantation and assisted reproductive technology, as well as the frequent medical monitoring which will be required of transplant subjects.

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01 (Estimated); Primary Completion 2018-07-24 (Actual); Study Completion 2018-07-24 (Actual)

PRIMARY OUTCOMES:
Successful Uterine Transplant | 2 years
  A successful uterine transplant surgery will be obtained by deceased-donor graft implantation and take (without rejection) and successful menstruation for a set period. Once stability is achieved, IVF will be performed and close monitoring of a pregnancy will be done. Finally, a successful healthy baby will be delivered via C-section. A successful uterine transplant will accomplish all the previously described metrics

CONTACTS AND LOCATIONS:
Overall Officials: Alexander T Maskin, MD, Principal Investigator — UNMC